CLINICAL TRIAL: NCT06754488
Title: A New Vesicocervical Urethral Reconstruction Technique Improves Urinary Continence in Patients After Laparoscopic Radical Prostatectomy: a Single-center Randomized Controlled Trial
Brief Title: A Technique Improves Urinary Continence in Patients Undergoing Laparoscopic Radical Prostatectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suzhou Municipal Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: K2024135K01
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-06

CONDITIONS: Posterior Bladder Wall Reconstruction; Anterior Bladder Wall Reconstruction; Anterior Bladder Wall Suspension
Keywords: prostate cancer; early urinary continence; laparoscopic radical prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Posterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- posterior reconstruction group (Experimental): In the posterior wall reconstruction group, laparoscopic radical prostatectomy was performed using an extraperitoneal approach:(1)The extraperitoneal space was established, and Trocar was placed.(2)The Retzius space was separated, the pelvic fascia on both sides of the prostate was incised, the bilateral puboprostatic ligaments were severed, and the dorsal vein complex (DVC) was sutured with 2-0 barb wire.(3)The bladder neck was severed.(4)The prostate and seminal vesicles were separated, the Denonvilliers fascia was opened, and the prostate gland was bluntly and sharply separated from the apex. The lateral prostatic ligaments were severed on both sides.(5)The prostate tip and urethra were severed.(6)Bladder neck reconstruction and bladder neck urethral anastomosis were performed: The bladder neck was reconstructed using the "inverted tennis racket" method to reduce the bladder neck, extend the back wall of the bladder, and anastomose the vesical-urethra.
  Interventions: Procedure: Posterior Reconstruction
- posterior reconstruction + anterior suspension group (Experimental): In the posterior reconstruction + anterior suspension group, laparoscopic radical prostatectomy with an extraperitoneal approach (steps 1 to 5) was performed similarly to the posterior wall reconstruction group.(6) The bladder neck was reconstructed using the "inverted tennis racket" method to reduce the bladder neck, extend the back wall of the bladder, and anastomose the vesical-urethra.(7)the anterior wall of the bladder was continuously sutured and fixed onto the muscular membrane of the lower margin of the symphysis pubis using a barb suture.
  Interventions: Procedure: Posterior Reconstruction; Procedure: anterior suspension
- Sham group (No Intervention): In the posterior reconstruction + anterior suspension group, laparoscopic radical prostatectomy with an extraperitoneal approach (steps 1 to 5) was performed similarly to the posterior wall reconstruction group.(6) The bladder neck was reconstructed using the "tennis racket" method to reduce the bladder neck, extend the back wall of the bladder, and anastomose the vesical-urethra.
- anterior suspension group (Experimental): In the posterior reconstruction + anterior suspension group, laparoscopic radical prostatectomy with an extraperitoneal approach (steps 1 to 5) was performed similarly to the posterior wall reconstruction group.(6) The bladder neck was reconstructed using the "tennis racket" method to reduce the bladder neck, extend the back wall of the bladder, and anastomose the vesical-urethra.(7)the anterior wall of the bladder was continuously sutured and fixed onto the muscular membrane of the lower margin of the symphysis pubis using a barb suture.
  Interventions: Procedure: anterior suspension

INTERVENTIONS:
Procedure: Posterior Reconstruction — Reconstruct the bladder neck using the "inverted tennis racket" method to narrow the bladder neck opening and lengthen the posterior bladder wall. Measure the length of the extended part.
  Arms: posterior reconstruction + anterior suspension group; posterior reconstruction group
Procedure: anterior suspension — The anterior wall of the bladder was continuously sutured and fixed onto the muscular membrane of the lower margin of the symphysis pubis using a 3-0 barb suture.
  Arms: anterior suspension group; posterior reconstruction + anterior suspension group

SUMMARY:
Laparoscopic radical prostatectomy (LRP) is the main treatment method for early prostate cancer, and postoperative urinary incontinence is one of the main complications after LRP. Urologists have applied various new operations in clinical practice to improve the urinary incontinence of patients after LRP surgery, but urinary incontinence is still the main problem affecting the quality of life of patients after surgery. In recent years, we have found that the new bladder neck urethral reconstruction method adopted by our department in LRP surgery can effectively improve the postoperative urinary incontinence of patients. In this study, a randomized controlled trial was intended to verify that the new bladder and neck urethral reconstruction technique could effectively improve early urinary control in patients after radical laparoscopic prostatectomy, and the patients were randomly divided into four groups by factorial design: posterior reconstruction group, posterior reconstruction +anterior suspension group, Sham group, and anterior suspension group to further verify the influencing factors of improved urinary control. The aim is to prove that the new operation can effectively reduce the urinary incontinence rate of patients after LRP, and analyze the mechanism of the new operation to improve the urinary incontinence of patients after LRP, and provide a new idea for the reconstruction of bladder neck and urethra during laparoscopic radical prostatectomy.

DETAILED DESCRIPTION:
Prostate cancer is a highly prevalent malignant tumor among men, ranking second in male malignant tumors. Radical prostatectomy (RP) is a primary treatment option for localized prostate cancer, with laparoscopic radical prostatectomy (LRP) being the most commonly used surgical method.

Currently, the evaluation of prostate surgery's effectiveness has expanded beyond merely improving patients' overall survival rates. Both doctors and patients now also prioritize the recovery of postoperative functions. Patel et al. proposed five consecutive criteria for evaluating RP outcomes:Long-term tumor control，Retention of urinary control function，Retention of erectile function，No surgical complications，Negative incisal margin.Urinary incontinence is a significant complication post-RP that severely impacts the quality of life and the willingness of patients to undergo RP. Thus, clinicians continuously improve surgical techniques to enhance urinary control post-RP.

Research indicates that retaining and reconstructing urinary control-related structures can influence postoperative urinary control. Despite various techniques being employed, there is no definitive evidence on the best method for postoperative urinary control. Current techniques to improve postoperative urinary incontinence include:Intraoperative retention of membranous urethra length (MUL)，Retention of bladder neck，Retention of neurovascular bundle (NVB)，Reconstruction of bladder neck.The internal urethral sphincter, located at the bladder neck, coordinates and controls urination. A study by Nyarangi-Dix et al. showed that preserving the bladder neck opening significantly improves urinary control post-LRP, with urinary control rates of 84.2%, 89.5%, and 94.7% at 3, 6, and 12 months, respectively. These rates were higher compared to those without bladder neck preservation, at 55.3%, 74.8%, and 81.4%.

The impact of NVB retention on urinary control remains controversial, but it may increase the positive resection margin rate. The external urethral sphincter also plays a crucial role in postoperative urine control.Some scholars found that maximizing the preservation of the membranous urethra during surgery improved urinary control rates at 30 days and 1 year post-surgery, reduced the use of urinary pads, and enhanced patients' quality of life.Various scholars have employed different reconstruction techniques to improve postoperative urinary control. For instance, ROCCO et al. used a posterior urethral fascia reconstruction technique, continuously suturing the severed ends of the anterior layer of Denonvilliers' fascia, the posterior bladder wall, the posterior wall of the external urethral sphincter, and the fibrous structure below the external urethral sphincter before vesical-urethral anastomosis. This technique restores the external urethral sphincter to its original anatomic position and reduces vesicourethral anastomosis tension.

The anterior suspension technique, first proposed by Walsh and later applied in LRP by Patel et al., involves suturing the dorsal vein complex (DVC) to the periosteum of the pubic arch to enhance anterior urethral wall support and restore elastic suspension. The Hood technique, another commonly used method, requires freeing the fat layer on the anterior bladder wall's surface to establish the surgical space without fully exposing the retropubic Retzius space. This preserves the suspension support structures around the retropubic urethra, ensuring its integrity.In China, Liu Zhibin et al. used anterior wall reconstruction and posterior wall strengthening techniques for bladder neck and urethra reconstruction to improve postoperative urine control.

These advancements in surgical techniques demonstrate the continuous effort to enhance the quality of life for prostate cancer patients undergoing radical prostatectomy by improving postoperative urinary control.

Even with the numerous surgical techniques available to improve postoperative urinary control for LRP patients, postoperative urinary incontinence remains a significant issue for many. In recent years, our center has adopted a novel bladder neck and urethra reconstruction method during laparoscopic radical prostatectomy for prostate cancer. We utilize the "inverted tennis racket" technique to reconstruct the bladder neck, which lengthens the posterior bladder wall, followed by vesicourethral anastomosis. Post-anastomosis, this is positioned at the upper margin of the symphysis pubis. The anterior bladder wall is then secured behind the symphysis pubis using a continuous 3-0 barb suture. This method has yielded improved results, significantly reducing the rate of postoperative urinary incontinence.

Prostate cancer patients admitted to the Department of Urology at Suzhou Hospital, affiliated with Nanjing Medical University, post-January 2025, were selected for the study. Eligible prostate cancer patients were randomly divided into four groups:1.Posterior wall reconstruction group,2.Posterior wall reconstruction + suspension group.3.Sham group.4.Anterior suspension group All four groups underwent laparoscopic radical prostatectomy via an extraperitoneal approach. During the bladder neck urethral reconstruction step, the experimental groups received the new bladder neck urethral reconstruction, while the control groups underwent conventional surgery. Patients were followed up post-surgery, comparing the urinary control status of both groups immediately after catheter removal and at 1 month, 3 months, 6 months, and 12 months post-surgery.

Inclusion Criteria:1.Age < 80 years old.2.Preoperative biopsy confirming prostate cancer.3.Clinical stages T1 and T2

Exclusion Criteria:

1.Diseases significantly increasing the risk of surgery or anesthesia (e.g., severe cardiovascular disease, respiratory disease, clotting disorders).2.Extensive bone or other organ metastases.3.History of urinary incontinence or transurethral resection of the prostate.4.Tumor invasion

Surgical Procedure for the Posterior Reconstruction Group:

(1)Establish the extraperitoneal space and place the Trocar.(2)Separate the Retzius space, incise the pelvic fascia on both sides of the prostate, sever the bilateral puboprostatic ligaments, and suture the dorsal vein complex (DVC) with 2-0 barb wire.(3)Treat the bladder neck: cut the anterior bladder neck wall sharply with an ultrasonic knife at the prostate-bladder neck junction (12 o'clock), revealing the posterior bladder neck wall. Separate the posterior bladder neck wall on both sides along the level between the bladder neck and prostate using an ultrasonic knife.Separate the prostate and seminal vesicles: find both vas deferens behind the bladder and cut them off, free both seminal vesicles, expose and cut off the lateral ligaments of the prostate with Hem-o-Lok. Open the Denonvilliers fascia and bluntly sharpen the prostatic gland to the apex.Cut off the prostate tip and urethra: cut the DVC with an ultrasonic knife, fully free the urethra at the prostate tip, preserving as much functional urethra length as possible. Cut the urethra with scissors, completely remove the prostate, and place it in a specimen bag without removing it from the body.Perform bladder neck reconstruction and bladder neck urethral anastomosis: reconstruct the bladder neck using the "inverted tennis racket" method to narrow the bladder neck opening and lengthen the posterior bladder wall. Measure the length of the extended part. Suture the bladder and urethra with a 2-0 sliding line from 5 o'clock, with a total of 8-10 stitches.This innovative method aims to improve postoperative urinary control and enhance the quality of life for patients undergoing laparoscopic radical prostatectomy.

Posterior Reconstruction + Anterior Suspension Group: Laparoscopic radical prostatectomy with an extraperitoneal approach (steps 1 to 5) was performed similarly to the posterior wall reconstruction group.(6) The bladder neck was reconstructed using the "inverted tennis racket" method to reduce the bladder neck, extend the back wall of the bladder, and anastomose the vesical-urethra.(7)the anterior wall of the bladder was continuously sutured and fixed onto the muscular membrane of the lower margin of the symphysis pubis using a barb suture.

Sham Group: Laparoscopic radical prostatectomy with an extraperitoneal approach (steps 1 to 5) was performed similarly to the posterior wall reconstruction group.(6) The bladder neck was reconstructed using the "tennis racket" method to reduce the bladder neck, extend the back wall of the bladder, and anastomose the vesical-urethra.

Anterior Suspension Group: Laparoscopic radical prostatectomy with an extraperitoneal approach (steps 1 to 5) was performed similarly to the posterior wall reconstruction group.(6) The bladder neck was reconstructed using the "tennis racket" method to reduce the bladder neck, extend the back wall of the bladder, and anastomose the vesical-urethra.(7)the anterior wall of the bladder was continuously sutured and fixed onto the muscular membrane of the lower margin of the symphysis pubis using a barb suture.

Assessment Methods for Urinary Incontinence: The primary assessment methods include the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF), daily urine pad usage, and 24-hour pad weight measurement. Post radical prostatectomy, the standard for urine control is achieved by either not using any urine pads or experiencing no urine leakage daily or by using only one safety urine pad. The ICIQ-SF and the 24-hour pad test were used to objectively evaluate urinary incontinence immediately after Foley catheter removal. Assessments were repeated at 1, 3, 6, and 12 months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

(1) Preoperative needle biopsy confirmed prostate cancer; (2) The clinical stage is T1 and T2

Exclusion Criteria:

(1) Diseases that significantly increase the risk of surgery or anesthesia, such as severe cardiovascular diseases, respiratory diseases, and coagulation disorders. (2) Patients with extensive bone metastasis or metastases to other organs (3) patients with a history of urinary incontinence and transurethral resection of the prostate. (4) Tumor invasion of bladder neck.

Max Age: 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The rate of continence | 1 month, 3 months, 6 months and 12 months after surgery
  Continence was defined as no more than 1 pads requirement daily by patients for normal physical activity and incontinence was defined as >1 pads daily.

CONTACTS AND LOCATIONS:
Locations (1):
- Suzhou Municipal Hospital, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sutherland DE, Linder B, Guzman AM, Hong M, Frazier HA 2nd, Engel JD, Bianco FJ Jr. Posterior rhabdosphincter reconstruction during robotic assisted radical prostatectomy: results from a phase II randomized clinical trial. J Urol. 2011 Apr;185(4):1262-7. doi: 10.1016/j.juro.2010.11.085. Epub 2011 Feb 22. PMID 21334025
- [Background] Soda T, Otsuka H, Koike S, Okada T. Baseline factors and surgical procedures affecting changes in lower urinary tract symptoms after robot-assisted radical prostatectomy: the impact of nerve-sparing. Int Urol Nephrol. 2024 Mar;56(3):989-997. doi: 10.1007/s11255-023-03859-9. Epub 2023 Oct 31. PMID 37907707
- [Background] Zhao X, Li K, Zhuang R, Liu H, He W, Dong W, Huang H, Huang J, Lin T. Comparison in Efficacy of Periurethral Reconstruction Leading to Urinary Continence Improvement After Robot-assisted Radical Prostatectomy. Ann Surg Oncol. 2024 Dec;31(13):8978-8985. doi: 10.1245/s10434-024-16225-5. Epub 2024 Sep 17. PMID 39287903
- [Background] Ortner G, Honis HR, Bohm J, Konschake M, Tokas T, Nagele U. Improved early continence following laparoscopic radical prostatectomy: the urethral hammock technique. World J Urol. 2024 Mar 16;42(1):168. doi: 10.1007/s00345-024-04857-x. PMID 38492077
- [Background] Sakai I, Harada K, Hara I, Eto H, Miyake H. Intussusception of the bladder neck does not promote early restoration to urinary continence after non-nerve-sparing radical retropubic prostatectomy. Int J Urol. 2005 Mar;12(3):275-9. doi: 10.1111/j.1442-2042.2005.01070.x. PMID 15828955
- [Background] Rocco F, Carmignani L, Acquati P, Gadda F, Dell'Orto P, Rocco B, Bozzini G, Gazzano G, Morabito A. Restoration of posterior aspect of rhabdosphincter shortens continence time after radical retropubic prostatectomy. J Urol. 2006 Jun;175(6):2201-6. doi: 10.1016/S0022-5347(06)00262-X. PMID 16697841
- [Background] Catarin MV, Manzano GM, Nobrega JA, Almeida FG, Srougi M, Bruschini H. The role of membranous urethral afferent autonomic innervation in the continence mechanism after nerve sparing radical prostatectomy: a clinical and prospective study. J Urol. 2008 Dec;180(6):2527-31. doi: 10.1016/j.juro.2008.08.020. Epub 2008 Oct 19. PMID 18930493
- [Background] Walz J, Burnett AL, Costello AJ, Eastham JA, Graefen M, Guillonneau B, Menon M, Montorsi F, Myers RP, Rocco B, Villers A. A critical analysis of the current knowledge of surgical anatomy related to optimization of cancer control and preservation of continence and erection in candidates for radical prostatectomy. Eur Urol. 2010 Feb;57(2):179-92. doi: 10.1016/j.eururo.2009.11.009. Epub 2009 Nov 11. PMID 19931974
- [Background] Harris MJ. The anatomic radical perineal prostatectomy: an outcomes-based evolution. Eur Urol. 2007 Jul;52(1):81-8. doi: 10.1016/j.eururo.2006.10.041. Epub 2006 Oct 30. PMID 17084506
- [Background] Walsh PC. Anatomic radical prostatectomy: evolution of the surgical technique. J Urol. 1998 Dec;160(6 Pt 2):2418-24. doi: 10.1097/00005392-199812020-00010. PMID 9817395
- [Background] Patel VR, Coelho RF, Palmer KJ, Rocco B. Periurethral suspension stitch during robot-assisted laparoscopic radical prostatectomy: description of the technique and continence outcomes. Eur Urol. 2009 Sep;56(3):472-8. doi: 10.1016/j.eururo.2009.06.007. Epub 2009 Jun 16. PMID 19560260
- [Background] Vis AN, van der Poel HG, Ruiter AEC, Hu JC, Tewari AK, Rocco B, Patel VR, Razdan S, Nieuwenhuijzen JA. Posterior, Anterior, and Periurethral Surgical Reconstruction of Urinary Continence Mechanisms in Robot-assisted Radical Prostatectomy: A Description and Video Compilation of Commonly Performed Surgical Techniques. Eur Urol. 2019 Dec;76(6):814-822. doi: 10.1016/j.eururo.2018.11.035. Epub 2018 Dec 2. PMID 30514568
- [Background] Walz J, Epstein JI, Ganzer R, Graefen M, Guazzoni G, Kaouk J, Menon M, Mottrie A, Myers RP, Patel V, Tewari A, Villers A, Artibani W. A Critical Analysis of the Current Knowledge of Surgical Anatomy of the Prostate Related to Optimisation of Cancer Control and Preservation of Continence and Erection in Candidates for Radical Prostatectomy: An Update. Eur Urol. 2016 Aug;70(2):301-11. doi: 10.1016/j.eururo.2016.01.026. Epub 2016 Feb 2. PMID 26850969
- [Background] Rocco B, Gregori A, Stener S, Santoro L, Bozzola A, Galli S, Knez R, Scieri F, Scaburri A, Gaboardi F. Posterior reconstruction of the rhabdosphincter allows a rapid recovery of continence after transperitoneal videolaparoscopic radical prostatectomy. Eur Urol. 2007 Apr;51(4):996-1003. doi: 10.1016/j.eururo.2006.10.014. Epub 2006 Oct 23. PMID 17079070
- [Background] Rocco B, Cozzi G, Spinelli MG, Coelho RF, Patel VR, Tewari A, Wiklund P, Graefen M, Mottrie A, Gaboardi F, Gill IS, Montorsi F, Artibani W, Rocco F. Posterior musculofascial reconstruction after radical prostatectomy: a systematic review of the literature. Eur Urol. 2012 Nov;62(5):779-90. doi: 10.1016/j.eururo.2012.05.041. Epub 2012 May 30. PMID 22664219
- [Background] Kim M, Park M, Pak S, Choi SK, Shim M, Song C, Ahn H. Integrity of the Urethral Sphincter Complex, Nerve-sparing, and Long-term Continence Status after Robotic-assisted Radical Prostatectomy. Eur Urol Focus. 2019 Sep;5(5):823-830. doi: 10.1016/j.euf.2018.04.021. PMID 29759661
- [Background] Dalela D, Jeong W, Prasad MA, Sood A, Abdollah F, Diaz M, Karabon P, Sammon J, Jamil M, Baize B, Simone A, Menon M. A Pragmatic Randomized Controlled Trial Examining the Impact of the Retzius-sparing Approach on Early Urinary Continence Recovery After Robot-assisted Radical Prostatectomy. Eur Urol. 2017 Nov;72(5):677-685. doi: 10.1016/j.eururo.2017.04.029. Epub 2017 May 6. PMID 28483330
- [Background] Egan J, Marhamati S, Carvalho FLF, Davis M, O'Neill J, Lee H, Lynch JH, Hankins RA, Hu JC, Kowalczyk KJ. Retzius-sparing Robot-assisted Radical Prostatectomy Leads to Durable Improvement in Urinary Function and Quality of Life Versus Standard Robot-assisted Radical Prostatectomy Without Compromise on Oncologic Efficacy: Single-surgeon Series and Step-by-step Guide. Eur Urol. 2021 Jun;79(6):839-857. doi: 10.1016/j.eururo.2020.05.010. Epub 2020 Jun 11. PMID 32536488
- [Background] Wagaskar VG, Mittal A, Sobotka S, Ratnani P, Lantz A, Falagario UG, Martini A, Dovey Z, Treacy PJ, Pathak P, Nair S, Roy B, Chakravarty D, Lewis S, Haines K 3rd, Wiklund P, Tewari A. Hood Technique for Robotic Radical Prostatectomy-Preserving Periurethral Anatomical Structures in the Space of Retzius and Sparing the Pouch of Douglas, Enabling Early Return of Continence Without Compromising Surgical Margin Rates. Eur Urol. 2021 Aug;80(2):213-221. doi: 10.1016/j.eururo.2020.09.044. Epub 2020 Oct 14. PMID 33067016
- [Background] Nyarangi-Dix JN, Radtke JP, Hadaschik B, Pahernik S, Hohenfellner M. Impact of complete bladder neck preservation on urinary continence, quality of life and surgical margins after radical prostatectomy: a randomized, controlled, single blind trial. J Urol. 2013 Mar;189(3):891-8. doi: 10.1016/j.juro.2012.09.082. Epub 2012 Sep 24. PMID 23017512